CLINICAL TRIAL: NCT00982384
Title: Comprehensive Disease Management Program in COPD Patients in the Community: Randomized Controlled Trial
Brief Title: Comprehensive Disease Management Program in Chronic Obstructive Pulmonary Disease (COPD) Patients in the Community
Acronym: COPD_CDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Ofra Kalter-Leibovici MD, Director of the Unit of Cardiovascular Epidemiology, Gertner Institute., Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHEBA-09-7120-OK-CTIL
Record Dates: First submitted 2009-09-14; First posted 2009-09-23 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease; Disease management; Pulmonary rehabilitation; Quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Disease Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disease management (Experimental): Comprehensive disease management in addition to best care according to clinical guidelines for COPD patients
  Interventions: Other: Disease management
- Best care (Active Comparator): Best care according to clinical guidelines for COPD patients
  Interventions: Other: Best care

INTERVENTIONS:
Other: Disease management — Disease management by COPD nurses, including active follow-up and coordination of care in addition to best care according to clinical guidelines for COPD patients
  Arms: Disease management
Other: Best care — Comprehensive care for COPD patients recommended in clinical guidelines
  Arms: Best care

SUMMARY:
The purpose of this study is to determine whether comprehensive disease management program combined with best care recommended in clinical guidelines, is more effective than best care alone in patients with advanced chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
The study objective is to evaluate the effectiveness of a comprehensive program among patients with advanced COPD, implemented by a multi-disciplinary team. The program consists of best care recommended in clinical guidelines, combined with disease management, compared to best care only.

The program will include designated COPD centers operated by multi-disciplinary teams (pulmonologists, nurse practitioners, physiotherapists, social workers and dietitians). Disease management will be provided in these centers by qualified designated nurses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 years or older
2. Advanced COPD

Exclusion Criteria:

1. Permanent tracheostomy
2. Heart failure with significant left-ventricular dysfunction
3. Severe other chronic disease
4. Significant cognitive impairment, Drug or alcohol abuse, inability to cooperate
5. No telephone or permanent address
6. Bedridden
7. Refusal to use telemonitoring equipment
8. Participation in another clinical trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1202 (Actual)
Dates: Start 2009-10; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Hospital admission for acute exacerbation of COPD or all-cause mortality | Within 2 to 5 years after randomization

SECONDARY OUTCOMES:
Total days of hospitalization for acute exacerbations of COPD | Within 2 to 5 years after randomization
Quality of life | Within 2 to 5 years after randomization
Total number of acute exacerbations of COPD | Within 2 to 5 years after randomization
Depression | Within 2 to 5 years after randomization
Functional capacity | Within 2 to 5 years after randomization
Spirometry parameters | Within 2 to 5 years after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ofra Kalter - Leibovici, M.D., Principal Investigator — Gertner Institute for Epidemiology & Health Policy Research, Sheba Medical Center; Gershon Fink, M.D., Study Director — Clalit Health Services
Locations (2):
- Israel (2):
  - Bat-Yam COPD Center, Bat Yam
  - COPD Center, Hadera, Hadera